CLINICAL TRIAL: NCT00344162
Title: A Familial Genetic Study on Preeclampsia: A Pilot Study
Brief Title: Family Study on Preeclampsia
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905097; 05-CH-N097
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-09-22

CONDITIONS: Preeclampsia
Keywords: Epidemiology; Population; Pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

SUMMARY:
This study will examine a possible genetic basis for preeclampsia, a disorder of high blood pressure and protein in the urine during pregnancy. Preeclampsia is a major pregnancy complication affecting both mother and baby. Previous research has shown that preeclampsia tends to run in certain families. This study will determine which genes may be involved in preeclampsia.

Women who have had preeclampsia (called the index woman) may be eligible for this study. They will be recruited through the Preeclampsia Foundation. In addition, the following relatives of the index woman may be enrolled:

* The child from the preeclampsic pregnancy
* The index woman's biological parents
* The index woman's siblings who have given birth or fathered a child and their family members

The study will exclude any index women or family members who have had chronic hypertension, diabetes, polycystic ovary syndrome, or whose pregnancy that involved preeclampsia was a multiple fetus pregnancy or that was conceived through use of fertility technology.

All women participants fill out a questionnaire to collect demographic data (e.g., age, race, marital status, etc.) and information on their medical and reproductive history, use of tobacco and medicines, and other factors that may be associated with preeclampsia syndrome. Women who have had preeclampsia or hypertension in pregnancy are asked to sign a medical record release form for study investigators to obtain a copy of the medical record for that pregnancy. All male and female participants provide a mouthwash rinse sample for extraction of DNA for gene studies. For babies too young to rinse with mouthwash, a soft brush is used to brush the inside of the mouth to collect cheek cells.

Mouthwash samples are analyzed for genes that may be associated with preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is a syndrome of hypertension accompanied by proteinuria. It is a major pregnancy complication, associated with premature delivery, fetal growth restriction, abruptio placentae, and fetal death, as well as maternal morbidity and mortality. Although preeclampsia has been recognized for centuries, the etiology of this disorder remains unknown. Familial clustering of preeclampsia has long been identified, leading to the concept of a genetic basis for this syndrome. We propose a familial genetic study of preeclampsia. As such a study is often difficult to do, we plan to conduct a pilot study to test the feasibility, logistics and examine frequency of genetic polymorphism of certain genes in the target population.

A total of 50 women who had preeclampsia during their first pregnancy will be identified through the Preeclampsia Foundation. Women who had chronic hypertension or diabetes prior to the first pregnancy will be excluded. We also will try to enroll their family members to this study. All subjects will be asked to complete a self-administered questionnaire and collect mouth wash samples. Women who reported having hypertension during pregnancy will be asked to sign a medical record release form. A copy of the medical record will be obtained to confirm the diagnosis of preeclampsia. DNA will be extracted from buccal cells. Frequency of polymorphisms for a number of candidate genes (e.g., HLA-G, AGT, eNOS, MTHFR, IL-1 beta, TNF-alpha, Prothrombin, and Factor V Leiden) will be examined. Information and experience gained from this pilot study will be most valuable for use to plan a main study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women who have had documented severe preeclampsia or eclampsia in their first pregnancy in the past 10 years will be potentially eligible for this study.

Through the index woman, we will invite her biological parents, siblings who have given birth or fathered a child and their family members to participate in this study.

EXCLUSION CRITERIA:

Excluded will be those who had chronic hypertension, diabetes, polycystic ovary syndrome, or the index pregnancy was a multifetal gestation or conceived by assisted reproductive technology.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-01-31; Study Completion 2006-09-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Boggess KA, Lieff S, Murtha AP, Moss K, Beck J, Offenbacher S. Maternal periodontal disease is associated with an increased risk for preeclampsia. Obstet Gynecol. 2003 Feb;101(2):227-31. doi: 10.1016/s0029-7844(02)02314-1. PMID 12576243